CLINICAL TRIAL: NCT04480957
Title: A Phase 1/2 Randomised, Double Blinded, Placebo Controlled, Ascending Dose Study to Assess the Safety, Tolerability, and Immunogenicity of ARCT-021 in Healthy Adult Subjects
Brief Title: Ascending Dose Study of Investigational SARS-CoV-2 Vaccine ARCT-021 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARCT-021-01
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Escalation Cohort dose 1 of ARCT-021, 21 - 55 years (Experimental): Escalation Cohort dose 1 of ARCT-021 administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose 1; Other: Placebo
- Escalation Cohort dose 2 of ARCT-021, 21 -55 years (Experimental): Escalation Cohort dose 2 of ARCT-021 administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose 2; Other: Placebo
- Escalation Cohort dose 3 of ARCT-021, 21 - 55 years (Experimental): Escalation Cohort dose 3 of ARCT-021 administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose 3; Other: Placebo
- Escalation Cohort dose 4 of ARCT-021, 21 - 55 years (Experimental): Escalation Cohort dose 4 of ARCT-021 administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose 4; Other: Placebo
- Expansion cohort dose regimen 1, 21 - 55 years. (Experimental): Expansion cohort dose regimen 1, administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose Regimen 1; Other: Placebo
- Expansion cohort dose regimen 2, 21 - 55 years. (Experimental): Expansion cohort dose regimen 2, administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose Regimen 2; Other: Placebo
- Expansion cohort dose regimen 1, 56 - 80 years (Experimental): Expansion cohort dose regimen 1, administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose Regimen 1; Other: Placebo
- Expansion cohort dose regimen 2, 56 - 80 years (Experimental): Expansion cohort dose regimen 2, administered through 0.5 mL intramuscular injection in the deltoid muscle.
  Interventions: Biological: ARCT-021 Dose Regimen 2; Other: Placebo

INTERVENTIONS:
Biological: ARCT-021 Dose 1 — ARCT-021 Dose 1 is an investigational vaccine comprising a self-replicating (replicon) mRNA that encodes for the full length spike protein of 2019-nCoV formulated in a lipid nanoparticle (LNP)
  Arms: Escalation Cohort dose 1 of ARCT-021, 21 - 55 years
Biological: ARCT-021 Dose 2 — ARCT-021 Dose 2 is an investigational vaccine comprising a self-replicating (replicon) mRNA that encodes for the full length spike protein of 2019-nCoV formulated in a lipid nanoparticle (LNP): ARCT-021
  Arms: Escalation Cohort dose 2 of ARCT-021, 21 -55 years
Biological: ARCT-021 Dose 3 — ARCT-021 Dose 3 is an investigational vaccine comprising a self-replicating (replicon) mRNA that encodes for the full length spike protein of 2019-nCoV formulated in a lipid nanoparticle (LNP): ARCT-021
  Arms: Escalation Cohort dose 3 of ARCT-021, 21 - 55 years
Biological: ARCT-021 Dose 4 — ARCT-021 Dose 4 is an investigational vaccine comprising a self-replicating (replicon) mRNA that encodes for the full length spike protein of 2019-nCoV formulated in a lipid nanoparticle (LNP): ARCT-021
  Arms: Escalation Cohort dose 4 of ARCT-021, 21 - 55 years
Biological: ARCT-021 Dose Regimen 1 — ARCT-021 dose regimen 1 is an investigational vaccine comprising a self-replicating (replicon) mRNA that encodes for the full length spike protein of 2019-nCoV formulated in a lipid nanoparticle (LNP): ARCT-021
  Arms: Expansion cohort dose regimen 1, 21 - 55 years.; Expansion cohort dose regimen 1, 56 - 80 years
Biological: ARCT-021 Dose Regimen 2 — ARCT-021 dose regimen 2 is an investigational vaccine comprising a self-replicating (replicon) mRNA that encodes for the full length spike protein of 2019-nCoV formulated in a lipid nanoparticle (LNP): ARCT-021
  Arms: Expansion cohort dose regimen 2, 21 - 55 years.; Expansion cohort dose regimen 2, 56 - 80 years
Other: Placebo — Sterile 0.9% saline

SUMMARY:
Determine safety and tolerability and immungenicity of investigational vaccine ARCT-021 in healthy adult volunteers.

DETAILED DESCRIPTION:
Randomized, double blinded (study site staff, subjects and Sponsor), placebo controlled, adaptive, ascending dose study evaluating administration of ARCT-021 in healthy adult subjects. 0.9% sterile saline will serve as a placebo control. Study drug (ARCT-021 or control) will be administered as an intramuscular (IM) injection. The study comprises two parts. In the Phase 1 part escalating dose levels given as a single injection to younger adults (21 to 55 years) will be evaluated sequentially. Two dose levels will be further evaluated in the Phase 2 part of the study in two expansion cohorts in younger adults (21 to 55 years) and in two elderly subject (56 to 80 years) cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged 21 to 80 at the time of informed consent.
2. Body Mass Index 18-35 kg/m2, inclusive, at screening
3. Willing to refrain from strenuous exercise/activity (for example heavy lifting, weight training, intense aerobics classes etc.) and alcohol for at least 72 hours prior to study visits
4. Temperature is less than 99.3 degrees Fahrenheit (37.4 degrees Celsius) at screening AND at the pre-dose evaluation on Day 1
5. Willing and able to comply with protocol-defined procedures and complete all study visits
6. Males must be surgically sterile or willing to use adequate contraception; females must be post-menopausal, surgically sterile or willing to use adequate contraception

Exclusion Criteria:

1. Pregnant or breast feeding
2. Clinically significant abnormalities in medical history
3. Out of range screening laboratory results
4. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
5. Uncontrolled hypertension (BP > 160/100 mm Hg)
6. Uncontrolled diabetes
7. Any history of autoimmune disease
8. Immunodeficiency of any cause
9. History of Chronic liver disease
10. Treatment with another investigational drug, biological agent, or device within one month of screening, or 5 half-lives of investigational drug, whichever is longer
11. Recent (within 1 year) history of, or current drug or alcohol abuse
12. Has any blood dyscrasias or significant disorder of coagulation
13. Has an acute illness, as determined by the investigator, with or without fever [temperature >38.0 degrees Celsius (100.4 degrees Fahrenheit)] within 72 hours prior to each vaccination
14. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
15. Received or plans to receive another vaccine within 4 weeks before study vaccination or at any time during the study.
16. Receipt of any other SARS CoV-2 or other experimental coronavirus vaccine at any time prior to study or planned during the study
17. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the Study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and dose-relationship of AEs | 56 days
  Safety and tolerability of ARCT-021 assessed by determining the incidence, severity and dose-relationship of AEs by dose

SECONDARY OUTCOMES:
Geometric mean titre for SARS-CoV-2-specific serum neutralizing antibody | Up to 56 days
  SARS-CoV-2-specific serum neutralizing antibody levels, expressed as GMT
Mean titre for SARS-CoV-2-specific serum neutralizing antibody levels | Up to 56 days
  SARS-CoV-2-specific serum neutralizing antibody levels, expressed as mean titer
Geometric mean fold rise in titre for SARS-CoV-2-spike protein specific neutralizing antibody levels | Up to 56 days
  GMFR in titre for SARS-CoV-2-spike protein specific neutralizing antibodies from before vaccination to each subsequent time point

OTHER OUTCOMES:
Increase in SARS-CoV-2--spike protein-specific binding antibody levels | Up to 56 days
  GMFR in SARS-CoV-2--spike protein-specific binding antibody levels from before vaccination to each subsequent time point
Geometric mean SARS-CoV-2--spike protein-specific binding antibody titre | Up to 56 days
  GMT for SARS-CoV-2--spike protein-specific binding antibody levels
Mean SARS-CoV-2--spike protein-specific binding antibody titre | Up to 56 days
  Mean titer for SARS-CoV-2--spike protein-specific binding antibody levels
SARS-CoV-2-specific serum neutralizing antibody seroconversion rate | 56 days
  Proportion of participants that are seronegative before vaccination achieving a titer of greater than or equal to 20 for SARS-CoV-2-specific serum neutralizing antibodies
SARS-CoV-2-specific serum neutralizing antibody seroconversion rate (seropositive baseline) | 56 days
  Proportion of participants that are seropositive before vaccination achieving a greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2-specific serum neutralizing antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low Guek Hong, MD, Principal Investigator — SingHealth Investigational Medicine Unit (IMU)
Locations (1):
- SingHealth Investigational Medicine Unit (IMU), Singapore General Hospital, Singapore, Singapore